CLINICAL TRIAL: NCT05034458
Title: Diet as Adjuvant Therapeutics in the Era of Biologics in Pediatric-onset Crohn's Disease.
Brief Title: Diet in Pediatric Crohn´s Disease Treated With Biologics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Principal Investigator, MARIA SOLEDAD ARCUCCI, principal investigator, Hospital Italiano de Buenos Aires
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5992
Record Dates: First submitted 2021-06-12; First posted 2021-09-05 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diet (Experimental): Patients will do biologic treatment according to international guidelines and will do Crohns Disease Exclusion Diet( modulen- phase one ant two CDED) for 12 weeks.They will be monitored periodically by interview and physical examination by physician and nutritionist, laboratory, fecal calprotectin.
  Interventions: Dietary Supplement: Crohn's disease exclusion diet
- Control (No Intervention): Patients with normal treatment( biologic treatment indicated for CD)

INTERVENTIONS:
Dietary Supplement: Crohn's disease exclusion diet — Patients will receive, in addition to their normal treatment, polymeric formula + diet
  Arms: Diet

SUMMARY:
Cded in remission patients with high calprotectin

DETAILED DESCRIPTION:
Due to the success of diet in achieving remission in mild-moderate forms of the disease, and an increasing number of patients with loss of response to available drugs despite increasing dose and pathophysiology of the disease, the aim of the present study is to evaluate whether there is response with the addition of diet therapy in patients with moderate/severe forms of CD receiving biologic therapy (infliximab or adalimumab) and presenting active disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients under 18 years of age
* With a diagnosis of CD
* Who have completed remission induction with biologic therapy
* Who are on maintenance biologic therapy
* Present calprotectin values higher than the limit values established by the laboratory (higher than 250 ug/g).

Exclusion Criteria:

* Children who are unable to receive enteral dietary intake
* Comorbidities affecting nutritional status and/or bone metabolism, growth or pubertal development
* Children already on special diets

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2021-05-14 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-20 (Actual)

PRIMARY OUTCOMES:
Number of Participants with calprotectin less than 250 at week 12 | week 12
  Number of participants who achieve normal fecal calprotectin after the diet
Level of calprotectin | week 12
  To evaluate the change of the calprotectin value at 0 and 12 weeks in patients with or without the addition of dietary therapy.

SECONDARY OUTCOMES:
Adherence | 12 weeks
  Number of patients that were able to continue the diet and not drop out during at least the 12 weeks of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Marina Orsi, M.D., Principal Investigator — Hospital Italiano
Locations (1):
- Hospital Italiano de Buenos Aires, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Arcucci MS, Menendez L, Orsi M, Gallo J, Guzman L, Busoni V, Lifschitz C. Role of adjuvant Crohn's disease exclusion diet plus enteral nutrition in asymptomatic pediatric Crohn's disease having biochemical activity: A randomized, pilot study. Indian J Gastroenterol. 2024 Feb;43(1):199-207. doi: 10.1007/s12664-023-01416-x. Epub 2023 Aug 23. PMID 37610564

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-05-13): https://cdn.clinicaltrials.gov/large-docs/58/NCT05034458/Prot_SAP_000.pdf
  • Informed Consent Form (2021-05-13): https://cdn.clinicaltrials.gov/large-docs/58/NCT05034458/ICF_001.pdf